CLINICAL TRIAL: NCT07367490
Title: Neuromuscular Electrical Stimulation Versus Electromyographic Biofeedback on Oropharyngeal Dysphagia in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayaa yousri hussien khalifa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/0059525
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuromuscular electrical stimulation + Selected physical therapy program (Experimental): It included 20 patients who received neuromuscular electrical stimulation using VitalStim Plus in addition to selected physical therapy program.
  Interventions: Device: Neuromuscular electrical stimulation; Other: Selected physical therapy program
- Electromyographic Biofeedback + Selected physical therapy program (Experimental): It included 20 patients who will receive electromyographic biofeedback in addition to selected physical therapy program.
  Interventions: Device: Electromyographic Biofeedback; Other: Selected physical therapy program
- Selected physical therapy program (Active Comparator): It included 20 patients who received selected physical therapy program only.
  Interventions: Other: Selected physical therapy program

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — Two pairs of electrodes were placed horizontally over the submental and paratracheal (thyroid cartilage) regions. Surged neuromuscular electrical stimulation was applied at a frequency of 80 Hz with a pulse duration of 200-300 µs. Stimulation was delivered for 30 minutes per session, five days per week, over an eight-week period.
  Arms: Neuromuscular electrical stimulation + Selected physical therapy program
Device: Electromyographic Biofeedback — It is a safe, simple, noninvasive treatment method means that can collect electromyographic signal of muscle activity for quantitative and qualitative analysis of neuromuscular functions.
  Other Names: EMG Biofeedback
  Arms: Electromyographic Biofeedback + Selected physical therapy program
Other: Selected physical therapy program — It includes lips exercise, tongue exercises, effortful swallowing maneuver, Mendelsohn maneuver and neck muscle exercise.
  Other Names: Physical therapy exercises

SUMMARY:
This study aims to investigate the effect of neuromuscular electrical stimulation versus electromyographic biofeedback on swallowing function and dysphagia severity in patients with stroke.

DETAILED DESCRIPTION:
Dysphagia is a common symptom seen in stroke patients, it is affected patients' nutrition supply, and may causes aspiration pneumonia. To solve the problem of nutritional support, nasogastric tubes are routinely indwelling to provide nutrition. This feeding method sometimes causes food reflux, aspiration, pneumonia, and discomfort and self-image acceptance.

Traditional exercise based on exercise like Shaker exercise, Chin resisted exercise and effortful training. Shaker exercise here is designed by professor Shaker has been regarded as popular rehabilitation training for dysphagia. Shaker exercise can strengthen upper esophageal sphincter, improving swallowing function.

Chin resisted exercise were developed to strengthen the suprahyoid muscles, whose contractions facilitate the opening of the upper esophageal sphincter, thereby improving bolus transfer.

Many studies reported that neuromuscular electrical stimulation can improve the swallowing function by enhancing swallowing coordination of post-stroke dysphagia patients. The improving of swallowing by surface electrical stimulation enhances raising and contraction of the hyoid bone of patients during swallowing. Neuromuscular electrical stimulation (VitalStim Plus), a method for stimulating muscles with short electrical pulses, is widely used in the therapy of stroke patients with pharyngeal dysphagia. It enhances the strength of the muscles associated with swallowing and facilitates reflex swallowing by sensory stimulation.

Using surface electromyography in post-stroke dysphagia cases increase ability of submental muscles activity and performance. Biofeedback or surface electromyography to ensure that target swallowing movements are being trained during rehabilitation, rather than maladaptive movements. Applying EMG-biofeedback add motivation to the therapy.

Both neuromuscular electrical stimulation and surface electromyography biofeedback improve recovery of swallowing function in stroke patients with dysphagia but yet there is no evidence about the most effective modality for improving swallowing in patients with acute stroke. So, this study was conducted to investigate and compare between effect of neuromuscular electrical stimulation and electromyographic biofeedback on swallowing function and dysphagia severity in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age were range from 45 to 60 years old.
* Presence of dysphagia from 3 weeks to 3 months, with preservation of cough reflex.
* Patients with severe moderate dysphagia according to dysphagia outcome and severity scale.
* Patients with sufficient cognitive abilities that enables them to understand and follow instructions.

Exclusion Criteria:

* Patients with distributed conscious level.
* Uncooperative patients.
* Patients with psychiatric disorders.
* Patients with syncope.
* Patients with dementia.
* Patients with history of dysphagia prior to onset of stroke.
* Patients with previous operation or injury in the neck.
* Patients with deficits in attention or cognition.
* Patients with cardiac pacemaker or history of seizures.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | 8 weeks
  The Functional Oral Intake Scale (FOIS) is a validated, seven-point observer-rated scale used to assess and monitor functional oral intake without increasing patient burden. Originally developed for individuals with neurogenic dysphagia, it demonstrates high reliability, interrater validity, and sensitivity to change. The scale ranges from level 1 (nothing by mouth) to level 7 (total oral diet with no restrictions) and is applied by trained observers to track eating abilities over time.
Dysphagia Outcome and Severity Scale (DOSS) | 8 weeks
  The Dysphagia Outcome and Severity Scale (DOSS) is an easy-to-administer, seven-point clinician-rated scale used to assess dysphagia severity and guide dietary and nutritional recommendations. It demonstrates strong intra- and interrater reliability and is based on objective parameters such as oral bolus transfer, pharyngeal residue, and airway protection. The scale ranges from level 1 (severe dysphagia with no safe oral intake) to level 7 (normal swallowing with no restrictions).

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ibrahim Rehab, PhD, Study Chair — Ass. Professor, Cairo University; Noura Abd Elhamid Elkafrawy, PhD, Study Director — Lecturer, Cairo University
Locations (1):
- Cairo University, Giza, Egypt